CLINICAL TRIAL: NCT01948076
Title: Use of a Pocket-sized Ultrasound Device as an Aid to the Physical Examination for Internal Medicine Residents
Brief Title: Evaluation of a Pocket-Sized Ultrasound Device As an Aid to the Physical Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Maria Yialamas, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011P-002845
Record Dates: First submitted 2013-09-16; First posted 2013-09-23 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-02

CONDITIONS: Splenomegaly; Pleural Effusion
Keywords: splenomegaly; pleural effusion
MeSH Terms: conditions — Splenomegaly; Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- resident without GE vscan (Placebo Comparator): baseline physical exam use
- resident with GE vscan (Active Comparator): residents with augmentation of physical exam by ultrasound
  Interventions: Device: resident with GE vscan

INTERVENTIONS:
Device: resident with GE vscan — resident with GE vscan
  Other Names: vscan
  Arms: resident with GE vscan

SUMMARY:
The 40 resident study subjects will be randomized to either receive a training session on use of a pocket-sized ultrasound or to receive training on physical exam skills. Following these sessions the subjects will have the opportunity to practice their skills during clinical rounds at BWH inpatient and outpatient settings. Four weeks after the training session all study subjects will take part in an assessment of their diagnostic skills. During this assessment they will be asked to complete an exam on a patient subject. Those randomized to the ultrasound group will be allowed to use their devices while the control group will use the traditional physical exam. Following the exams, resident study subjects will be asked to indicate whether they detected any of the following abnormalities on their exams: pleural effusion, hepatomegaly, cirrhotic liver, splenomegaly, ascites, aortic stenosis, mitral regurgitation, right atrial pressure, abdominal aortic aneurysm, deep vein thrombosis. Resident study subjects will also complete a questionnaire about the physical exam and use of the ultrasound. Prior to the assessment, all patients will undergo ultrasound by an attending radiologist, and these results will serve as the "gold standard" for our study.

DETAILED DESCRIPTION:
II. Specific Aims:

Study population: Internal medicine residents at an academic center

Patient population: A broad population of patients with diverse clinical conditions including cardiac and vascular disease, malignancy, rheumatologic disease, liver disease, renal failure, and others. This population will reflect the diversity of patients seen by internal medicine residents during their training.

Physical findings being studied:

1. Abdominal: hepatomegaly, cirrhotic liver, splenomegaly, ascites, abdominal aortic aneurysm
2. Lungs: pleural effusion, pneumothorax, paralyzed hemidiaphragm.
3. Cardiac: pericardial effusion, mitral regurgitation, tricuspid regurgitation, aortic insufficiency, aortic stenosis, right atrial pressure.

Primary Aim:

Determine the diagnostic accuracy of residents using a pocket-sized ultrasound device compared with residents using more traditional physical exam techniques for the physical findings mentioned above.

Secondary Aims:

* Determine whether medicine residents improve their physical exam diagnostic skills after receiving training with pocket-sized ultrasound devices.
* Determine the additional diagnostic benefit of pocket-sized ultrasound versus a traditional physical exam.
* Assess the diagnostic physical exam skills of medicine residents as compared with expert diagnosticians.
* Assess the diagnostic ultrasound skills of medicine residents as compared with trained radiologists using pocket-sized ultrasounds.
* Assess the degree of agreement between expert physical diagnosticians and trained radiologists using pocket-sized ultrasound.
* Evaluate the ability of residents to integrate ultrasound examination into their daily patient care routines

III. Subject Selection:

Inclusion Criteria:

All interns and residents in the BWH internal medicine residency program who responded to a recruitment email and agreed to participate.

Exclusion Criteria:

* Radiology Preliminary residents
* Residents with previous formalized ultrasound training that included a practical component

Resident Recruitment Methods:

All interns and residents in the BWH internal medicine residency program will be invited to participate in the study. The study will be advertised via email and announcements at residency educational conferences. Because Dr. Katz and Dr. Yialamas are part of the BWH residency leadership, they will not participate in the recruitment of residents to avoid a potential undue pressure to participate.

Patient Recruitment Methods:

Advertisements will be sent to selected faculty within the departments of medicine and radiology with details of patient involvement and the selected physical findings which will be studied. Patients will be asked by their treating physician or radiologist involved in their care if they can be contacted by the study coordinator. The coordinator will then assess interest and availability. Patients will then be consented if they agree to participate. Fourteen patient-subjects will ultimately be selected to participate in our assessment program. They will be compensated $350 for participating.

IV. Subject Enrollment

Forty of the residents who responded to the email advertisement will be randomly selected to be enrolled. Each resident enrolled will be consented by one of the investigators prior to participating in the study. The verbal consent process will assure subjects that study data and results will not appear in their residency record, or be used in any way by the residency program. They will therefore remain wholly within the purview of the investigation staff, and will not form any part of their residency evaluation. Each of the forty residents who participates in our study will receive a compensation of $150 for their time.

V. Study Procedures

Randomization and Curricular Training The 40 participating residents will be randomized to either the control or intervention group by having them blindly pick small pieces of paper with numbers out of a paper bag. All residents will participate in a 2 hour physical exam education session led by senior internal medicine faculty. Those randomized to the ultrasound group will also attend a 2 hour pocket-ultrasound training session which will be run by a BWH faculty radiologist and a BWH faculty echocardiographer. Following this training session, each of the 20 residents will be given a pocket-sized ultrasound device which they will be able to use as an adjunct to their physical exam while in clinic or on inpatient wards. Because the resident physicians are not trained ultrasound radiologists, these ultrasound studies will be informal and the results will not become part of any patient's medical record. Participants in the control arm of the study will not receive pocket-sized ultrasound devices nor will they receive training on how to use the machines.

Physical Exam Assessment Session Four weeks after randomization, all 40 of the resident subjects will attend a half-day physical exam assessment. This assessment will take place in the Brigham Circle Medical Associates Clinic on the Third Floor of the BWH Shapiro Cardiovascular Building. The assessment will also include the participation of 14 patient subjects who will be recruited ahead of time.

At the start of the day, each of the 14 patient subjects will be examined by two senior internal medicine clinicians to determine the presence of the physical exam findings being studied. Each patient subject will also undergo ultrasound evaluation by two BWH radiologists or echocardiographers to radiographically confirm the presence of the abovementioned physical findings. The "gold standard" for this study will be clinically detectable physical findings (as confirmed by senior clinicians) that are also confirmed by an ultrasound study performed by a radiologist or echocardiographer.

Patient study subjects will each be assigned to a clinic room and study subjects will rotate through each of the 14 rooms over the course of the half-day session. Each interaction will last 5 minutes and will consist of a focused physical examination of the patient. All 40 medicine residents will perform a routine physical exam on each patient and will document their findings. The 20 residents in the intervention group will also perform an exam on the same patients using a pocket-sized ultrasound and will document their findings.

Following the assessment, those study subjects randomized to the control group will have the opportunity to participate in a brief ultrasound training session, and they will also have a chance to practice using the ultrasounds during clinical practice over the following week.

VI. Biostatistical Analysis

Data collected during the assessment will include both binary variables for the presence of the aforementioned physical exam findings as well as to categorize the severity of each finding (mild, moderate, severe). Clinical definitions for these categories will be defined ahead of time. In addition, a short questionnaire will be distributed to all of the subjects and patient study subjects. The questionnaire will ask subjects about their comfort in performing various aspects of the physical exam, their use of handheld ultrasound devices, as well as their experiences teaching medical students and residents the physical exam. Patient study subjects will answer a questionnaire about their attitude towards being examined by a physician using a handheld ultrasound device.

Primary outcome measure: Physical exam diagnostic accuracy of residents compared with the diagnostic accuracy of residents using pocket-sized ultrasound devices.

Secondary outcome measures:

1. For the sub-group of residents with pocket-sized ultrasounds: comparing the diagnostic accuracy of routine physical exam versus with the ultrasound (i.e. how much additional diagnostic yield did the ultrasound provide?).
2. Comparing the diagnostic accuracy of physical exams by medical residents with the exams performed by the expert clinicians.
3. Comparing the diagnostic accuracy of pocket-sized ultrasounds performed by medical residents with the studies performed by expert radiologists and echocardiographers.
4. Assess the degree of agreement between expert physical diagnosticians and trained radiologists using pocket-sized ultrasound.

VII. Risks and Discomforts

We see no potential for harm to either study subjects or patient study subjects in this study. Ultrasound is a safe modality that does not involve ionizing radiation. We do not anticipate any pain or discomfort to our patient study subjects.

If any previously-unknown abnormalities are noted by our faculty radiologists or study subjects while performing an ultrasound on patient study subjects, the patient's primary care physician will be notified.

VIII. Potential Benefits The benefits of our study for participants will be the satisfaction of participating in a research study that has the potential to ultimately improve patient care.

We believe the potential global benefits from our study are significant. If handheld ultrasound devices prove to be helpful to internal medical residents in their physical assessment of patients, we would recommend that these machines be made available through the residency program. We hypothesize that handheld ultrasounds will enable internists to augment their physical exam skills with a direct impact on improving patient care.

IX. Monitoring and Quality Assurance

Because our study does not involve any potential harm to participants we do not anticipate the need for an independent safety monitoring board. All participants will, however, be encouraged to report any possible adverse events to our study coordinator, and participants will have the option of withdrawing from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* All interns and residents in the BWH internal medicine residency program who responded to a recruitment email and agreed to participate.

Exclusion Criteria:

* • Radiology Preliminary residents

  * Residents with previous formalized ultrasound training that included a practical component

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Yialamas, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ojeda JC, Colbert JA, Lin X, McMahon GT, Doubilet PM, Benson CB, Wu J, Katz JT, Yialamas MA. Pocket-sized ultrasound as an aid to physical diagnosis for internal medicine residents: a randomized trial. J Gen Intern Med. 2015 Feb;30(2):199-206. doi: 10.1007/s11606-014-3086-4. Epub 2014 Nov 12. PMID 25387438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning in Septemeber 2012 all internal medicine residents at Brigham and Women's hospital were invited to participate and the first 40 residents to respond to email advertisement were enrolled.
Pre-assignment Details: Residents with formal ultrasound training were to be excluded but none of the potential participants had had formal training.
Groups:
- Control Group: Performed only physical exam with no access to ultrasoun
- Intervention Group: Received training and access to ultrasounds. During assessment performed physical exam first followed by ultrasound exam
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resident Without GE Vscan | Resident With GE Vscan | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (2.3) | 29.5 (1.9) | 29.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Diagnostic Ability of the Intervention Group's Ultrasound Exam to the Control Group's Physical Exam
Description: The primary outcome is a comparison of the diagnostic ability of the intervention group as recorded after performing an ultrasound exam and the control group using traditional physical examination techniques. We compared the two groups using the average physical findings correctly identified as present or absent as reflected by a "Present Score" (average # of findings identified out of 17 possible findings) and "Absent Score" (average # of findings identified out of 95 possible). The former is a gauge of a resident's ability to correctly identify present abnormalities while the latter is an assessment of correctly identifying a normal examination when findings are absent. The residents used a examination form to indicate whether or not they felt the physical abnormality was present or absent and how confident he or she was in their answer. This was compared with the gold standard which was presence or absence of the abnormality on professional ultrasound.
Time Frame: one month
Population: All residents were analyzed. There was one withdrawal due to family emergency
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Resident Without GE Vscan | Resident With GE Vscan
Number analyzed (Participants) | 20 | 19
units on a scale
  Present Score | 6.4 [5 to 8] | 7.6 [5 to 9]
  Absent Score | 79.6 [74.5 to 84.5] | 79.3 [78 to 86]
Statistical Analysis 1: Comparison: Resident Without GE Vscan vs Resident With GE Vscan; Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Improvement in Diagnostic Ability Within the Intervention Group
Description: For the secondary outcome, we assessed whether there was an improvement in the diagnostic ability of those in the intervention group using traditional physical examination techniques as compared to using the ultrasound device. We compared the two arms using the average physical findings correctly identified as present or absent as reflected by a "Present Score" (average # of findings identified out of 17 possible findings) and "Absent Score" (average # of findings identified out of 95 possible). The residents used a examination form to indicate whether or not they felt the physical abnormality was present or absent using their physical exam alone and then again after using the ultrasound. This was compared with the gold standard which was presence or absence of the abnormality on professional ultrasound.
Time Frame: one month
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Groups:
- Intervention Group (Using Physical Exam Only): Baseline physical exam prior to using the ultrasound
- Intervention Group (Using Ultrasound): residents with augmentation of physical exam by ultrasound
Arm/Group | Intervention Group (Using Physical Exam Only) | Intervention Group (Using Ultrasound)
Number analyzed (Participants) | 19 | 19
units on a scale
  Present Score | 6.7 [5 to 9] | 7.6 [5 to 9]
  Absent Score | 79.3 [78 to 86] | 79.1 [78 to 87]
Statistical Analysis 1: Comparison: Intervention Group (Using Physical Exam Only) vs Intervention Group (Using Ultrasound); Test type: Superiority or Other; p = 0.043, McNemar

ADVERSE EVENTS:
Arm/Group | Resident Without GE Vscan | Resident With GE Vscan
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes